CLINICAL TRIAL: NCT07221513
Title: A Phase 2a, Open-Label Study to Assess the Safety, Tolerability, and Efficacy of JK07 in Participants With Heart Failure and Group 2 Combined Post-Capillary and Pre-Capillary Pulmonary Hypertension (RENEU-PH)
Brief Title: Study of JK07 in Patients With Heart Failure and WHO Group 2 Combined Post- and Pre-Capillary Pulmonary Hypertension
Acronym: RENEU-PH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Salubris Biotherapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JK07.2.04
Record Dates: First submitted 2025-08-20; First posted 2025-10-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HFrEF - Heart Failure With Reduced Ejection Fraction; HFpEF - Heart Failure With Preserved Ejection Fraction; Group 2 Pulmonary Hypertension
Keywords: Heart Failure; Heart Failure with Reduced Ejection Fraction; HFrEF; HFpEF; Heart Failure with Preserved Ejection Fraction; Group 2 Pulmonary Hypertension; Pulmonary Hypertension; cpcPH; Heart Failure NYHA Class III; Heart Failure NYHA Class II; Systolic Heart Failure; Diastolic Heart Failure; Neuregulin 1; NRG-1; ErbB4; HER3; HER4
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary; Heart Failure, Systolic; Heart Failure, Diastolic; Fibromatosis, Gingival, 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JK07 high dose (Experimental): JK07 administered by intravenous (IV) infusion
  Interventions: Drug: JK07

INTERVENTIONS:
Drug: JK07 — JK07 is a fully human anti-human epidermal growth factor receptor 3 (also known as ErbB3 or HER3) antibody fused with the epidermal growth factor (EGF)-domain of Neuregulin (NRG)-1b protein.

SUMMARY:
This is a Phase 2a, open-label, multiple-dose study to assess the safety, tolerability, and efficacy of JK07 in participants 18 to 85 years of age with diagnosed HF and cpcPH.

At least 20 and up to approximately 30 participants will be enrolled and receive JK07 high dose in this open-label trial.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with HF New York Heart Association Class II-III.
* Participants will be classified as having HFrEF (LVEF ≤ 40%) or HFpEF (LVEF >40% and ≤70%).
* Right heart catheterization (RHC) based evidence of cpcPH:
* PVR ≥2.5 WU; AND
* mPAP ≥25 mmHg; AND
* PAWP ≥16 mmHg

Key Exclusion Criteria:

* Diagnosis of PH in World Health Organization (WHO) Group 1, WHO Group 3, WHO Group 4, or WHO Group 5.
* Contraindicated to RHC that can be left in place for approximately 6 hours.
* A diagnosis of pre-existing lung disease including congenital abnormalities, full or partial pneumonectomy, or previous therapeutic radiation of lungs or mediastinum.
* Body mass index (BMI) >45 kg/m² at screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of TEAEs [Safety and tolerability] | Study entry through week 26
  Incidence and severity of treatment emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetic - Cmax | Study entry through week 26
  Characterize the JK07 PK profile through Peak Plasma Concentration (Cmax) following IV administration
Pharmacokinetics - Tmax | Study entry through week 26
  Characterize the JK07 PK profile through Time to Peak Plasma Concentration (Tmax) following IV administration
Pharmacokinetics - AUC0-last | Study entry through week 26
  Characterize the JK07 PK profile through area under the concentration-time curve from time 0 to last quantifiable concentration (AUC0-last) following IV administration
Pharmacokinetics - AUC0-inf | Study entry through week 26
  Characterize the JK07 PK profile through area under the concentration-time curve from time 0 to infinity (AUC0-inf) following IV administration
Pharmacokinetics - t1/2 | Study entry through week 26
  Characterize the JK07 PK profile through half-life (t1/2) following IV administration
Pharmacokinetics - λz | Study entry through week 26
  Characterize the JK07 PK profile through elimination rate constant (λz) following IV administration
Pharmacokinetics - CL | Study entry through week 26
  Characterize the JK07 PK profile through systemic clearance (CL) following IV administration
Pharmacokinetics - Vz | Study entry through week 26
  Characterize the JK07 PK profile through volume of distribution (Vz) following IV administration

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Francis Heart and Vascular Institute, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No